CLINICAL TRIAL: NCT01629459
Title: Effects of Resistance Exercise Training on Cardiac, Metabolic and Muscle Function and Quality of Life in Barth Syndrome
Brief Title: Resistance Exercise in Barth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201205024
Record Dates: First submitted 2012-06-20; First posted 2012-06-27 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Barth Syndrome
Keywords: exercise; strength; training; barth syndrome; mitochondria; amino acid; protein
MeSH Terms: conditions — Barth Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Resistance exercise training
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistance exercise training (Experimental): Participants will undergo resistance exercise training 3x/wk for 12 weeks at a physical therapy or cardiac rehabilitation facility near the participant's home.
  Interventions: Behavioral: Resistance exercise and protein supplementation

INTERVENTIONS:
Behavioral: Resistance exercise and protein supplementation — Resistance exercise training will occur 3x/wk for 12 wks at a physical therapy or cardiac rehabilitation facility near the participant's home. Participant will take 42 grams of supplementation protein daily.

SUMMARY:
Barth syndrome (BTHS) is a disorder that is characterized by heart failure, exercise intolerance and skeletal muscle weakness. Preliminary evidence demonstrates that endurance exercise training does not significantly improve exercise tolerance in BTHS. Because endurance exercise training targets a metabolic pathway that is adversely affected by BTHS, the investigators hypothesized that resistance training may improve exercise tolerance in BTHS because this type of training targets a different metabolic pathway than does endurance exercise. Therefore, the overall objective of the pilot/feasibility/proof-of-concept proposal is to collect preliminary data on the following hypothesis: Supervised resistance exercise training (3x/wk, 45min, 12 wks) will improve exercise tolerance, heart function, muscle strength and quality of life, and will be found safe in adolescents and young adults with BTHS.

DETAILED DESCRIPTION:
Barth syndrome (BTHS) is an X-linked disorder characterized by severe mitochondrial dysfunction, cardiomyopathy, skeletal muscle weakness and exercise intolerance. Preliminary evidence from our group has demonstrated that a 12-week endurance (i.e. aerobic) exercise training program increases exercise tolerance only modestly (~5%) in participants with BTHS with no effect on heart or skeletal muscle function. Other populations, including non-BTHS heart failure, appear to receive a greater benefit from endurance exercise training (e.g. ~15-25% increase in exercise tolerance) than does BTHS. The blunted effect of endurance exercise training in BTHS may be due to the inherent pathogenesis of BTHS: genetic mitochondrial dysfunction in type I (oxidative>glycolytic capacity) muscle fibers. Endurance exercise training typically results in increased mitochondrial density and enzyme function (primarily in type I muscle fibers) in other populations; however, in BTHS, due to maternally inherited mitochondrial dysfunction, endurance exercise training may result in the generation of more impaired mitochondria thus limiting any beneficial effect of endurance training on exercise tolerance. Thus, it may be more beneficial to target type II (glycolytic>oxidative capacity) muscle fibers with exercise training when attempting to increase exercise tolerance in BTHS. Indeed, previous evidence from non-BTHS heart failure has shown that resistance exercise training (RET) increases exercise tolerance, skeletal muscle strength, and heart function and improves quality of life in these individuals. Currently it is unknown if RET is effective in improving these variables in those with BTHS and is the focus of this proposal. Establishing the safety and efficacy of RET in BTHS could lead to clinical recommendations of regular RET instead of or in combination with endurance exercise training for the standard of care treatment of individuals with BTHS. Therefore, the overall objective of the pilot/feasibility/proof-of-concept proposal is to collect preliminary data on the following hypothesis: Supervised RET (3x/wk, 45min, 12 wks) with diet standardization (meeting at least minimum RDA recommendations for adolescents/young adults- 52-56 g protein/day) and protein supplementation (whey protein isolate, 42 g/day, Unjury Medical Quality Protein, Reston, VA ) will improve exercise tolerance, left ventricular function, muscle strength and quality of life, and will be found safe in adolescents and young adults with BTHS. In addition, our preliminary data suggest there is impaired protein metabolism and skeletal muscle atrophy in BTHS. Typically, in other populations, whole-body and skeletal muscle protein synthesis increases with RET; however, this is unclear in BTHS. Thus, as a secondary aim, we will examine the effect of RET on whole-body protein metabolism in BTHS. We aim to address these hypotheses through left ventricular function, skeletal muscle strength, body composition, exercise tolerance, and whole-body protein metabolism measurements at baseline and following a 3 month supervised RET program in 3 participants with BTHS (ages 15-30 yrs). Supervised RET programs will be uniformly designed, but individualized and performed at a physical therapy or cardiac rehabilitation facility near the participant's home. Protein supplementation (whey protein isolate, 42 g/day) will be ingested by the participants in conjunction with the RET program. Nutritional status will be evaluated at baseline, mid-training (6-weeks) and post-training through plasma levels of pre-albumin and amino acid profile. Left ventricular function will be examined using 2-D, Doppler and tissue Doppler echocardiography, skeletal muscle strength will be measured using isotonic and isokinetic dynamometry, body composition using dual energy x-ray absorptiometry, exercise tolerance will be measured using graded exercise testing and indirect calorimetry, whole-body protein metabolism by stable-isotope tracer methodology and mass spectrometry, and quality of life will be measured by the Minnesota Living with Heart Failure Questionnaire. We expect to find that RET is safe in BTHS, and effectively improves cardiac function, skeletal muscle strength and mass, whole-body protein synthesis and quality of life. Preliminary data from this proposal will be used in larger federal or association grant applications examining the cardiovascular, musculoskeletal and protein metabolic effects of RET in BTHS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-35 years
2. Sedentary (exercises less than 2x/wk)
3. Motivated to exercise (BTHS only)
4. Stable on medications for ≥ 3 months (BTHS only)
5. Lives in North America
6. Lives in the St. Louis area (Controls only)

Exclusion Criteria:

1. Unstable heart disease
2. Cardiac transplantation

Ages: 15 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in exercise tolerance | Enrollment, 3 months
  This study will examine the effect of resistance exercise training on exercise tolerance: peak oxygen consumption, exercise time and exercise work during graded exercise test on cycle ergometer

SECONDARY OUTCOMES:
Change in muscle strength | Enrollment, 3 months
  This study will measure the effect of resistance exercise training on muscle strength measured by 1-repetition maxium testing on universal equipment
Change in quality of life | Enrollment, 3 months
  This study will examine the effect of resistance exercise training on quality of life measures by Minnesota living with heart failure questionnaire
Change in left ventricular systolic strain | Enrollment, 3 months
  This study will examine the effect of resistance exercise training on left ventricular systolic strain measured by tissue Doppler echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No